CLINICAL TRIAL: NCT05634954
Title: A Phase 1 Study to Assess the Safety, Radiation Dosimetry and Biodistribution, and Basic Pharmacokinetics of [18F]GEH121224 and Determine the Optimal Timing of Imaging in Patients With Locally Advanced or Metastatic Breast Cancer.
Brief Title: Study to Evaluate Safety and Dosimetry of [18F]GEH121224 in Patients With Locally Advanced or Metastatic Breast Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Business Decision
Sponsor: GE Healthcare (Industry)
Collaborators: Laboratory Corporation of America (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: GE-226-004
Record Dates: First submitted 2022-11-22; First posted 2022-12-02 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer
Keywords: HER2 positive; Breast Oncology
MeSH Terms: conditions — Breast Neoplasms | interventions — Injections

STUDY DESIGN:
Intervention Model Description: Patients will be enrolled into 1 of 2 groups in a sequential manner. Group 1 will allow to study [18F]GEH121224 Biodistribution and Radiation Dosimetry. Group 2 will allow to study [18F]GEH121224 PET/CT Scan Test Retest.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- [18F]GEH121224 - Group 1 - Biodistribution (Experimental)
  Interventions: Drug: GEH121224 (18F) Injection; Diagnostic Test: Dynamic and Static - PET/CT Scan
- [18F]GEH121224 - Group 2 - Reproducibility (Experimental)
  Interventions: Drug: GEH121224 (18F) Injection; Diagnostic Test: Static - PET/CT Scan

INTERVENTIONS:
Drug: GEH121224 (18F) Injection — Single GEH121224 (18F) Injection
Diagnostic Test: Dynamic and Static - PET/CT Scan — Group 1: Dynamic whole-body PET/CT scan will start at the time of injection (8 sequential scans over 90 minutes anticipated) followed by static whole-body scans starting at 120 minutes and 240 minutes after injection.
  Arms: [18F]GEH121224 - Group 1 - Biodistribution
Diagnostic Test: Static - PET/CT Scan — Group 2: Static whole-body scans
  Arms: [18F]GEH121224 - Group 2 - Reproducibility

SUMMARY:
The study described in this protocol is a Phase 1, single center clinical trial to evaluate the safety and potential of [18F]GEH121224 as a PET radiotracer for the diagnostic imaging of HER2 positive breast cancer lesions. A group of 6 patients will be selected to perform a dosimetry study with [18F]GEH121224 followed by another group of 6 patients in a test-retest study. The results of this study will provide crucial information to guide the development of [18F]GEH121224 for the detection of HER2 status in advanced breast cancer patients. This study will use established methods for characterizing the radiation dosimetry, biodistribution and basic pharmacokinetics of a radiotracer.

DETAILED DESCRIPTION:
Group 1 : Six female patients with locally advanced or metastatic breast cancer and with HER2-positive primary tumor status will be included. These patients will receive a single injection of GEH121224 (18F) Injection and will then undergo a dynamic whole-body PET/CT scan starting at the time of injection (8 sequential scans over 90 minutes anticipated) followed by static whole-body scans starting at 120 minutes and 240 minutes after injection. Blood samples will be collected at specified time points during imaging for pharmacokinetic analysis. Safety and imaging data will be reviewed on an ongoing basis after dosing of each patient in Group 1. The injected activity may be adjusted for subsequent patients in Group 1 based on this review. A complete aggregate review of safety and imaging data will be performed by the Sponsor once all 6 patients in Group 1 have been dosed. If no safety concerns are raised, enrollment into Group 2 will start. The injected radioactivity may also be optimized before enrolling patients in Group 2. Review of safety data is described in the Safety Data Review Plan.

Group 2 : Six female patients with locally advanced or metastatic breast cancer and with HER2-positive primary tumor status will be included in Group 2 and will receive a single injection of GEH121224 (18F) Injection on each of 2 separate days. On Imaging Day 1, patients will receive a single injection of GEH121224 (18F) Injection and will then undergo [18F]GEH121224 PET imaging at the optimal scan time identified in Group 1. Within 3 weeks (3 to 21 days; Imaging Day 2), patients will receive a second single injection of GEH121224 (18F) Injection and again undergo [18F]GEH121224 PET imaging at the optimal scan time identified in Group 1.

Patient safety will be monitored throughout the course of the study, including a 24-hour safety follow-up by phone after each dose of [18F]GEH121224.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged ≥18 years
* Willingness and ability to comply with study procedures and signed and dated informed consent
* For women of child-bearing potential, negative urine pregnancy test at screening and o on the day of investigational medicinal product (IMP) administration (with the result known before IMP administration) and willingness to use contraception (barrier, abstinence, non-hormonal) for 3 weeks after injection of [18F]GEH121224
* Life expectancy >3 months
* Diagnosis of locally advanced or metastatic breast cancer
* Target lesion diameter of ≥15 mm that has not been previously treated with radiotherapy
* Histologically confirmed locally advanced/metastatic breast cancer with a biopsy within the past 12 months confirming HER2-positive status by either IHC or FISH from primary tumor
* Previously received no more than 1 prior lines of systemic chemotherapy (including anti HER2 therapy) for metastatic breast cancer
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
* Adequate organ function as defined by:

Hemoglobin ≥10 g/dL White blood cell count ≥3.0 × 109/L Platelet count ≥75 × 109/L Serum creatinine ≤1.4 mg/dL Aspartate aminotransferase and alanine aminotransferase ≤2× upper limit of normal (ULN) Total bilirubin ≤2× ULN or 3.0 mg/dL in patients with Gilbert's syndrome

* At least one lesion is fluorodeoxyglucose (FDG)-avid

Exclusion Criteria:

* Patient has a primary non-breast malignancy (small dermatological malignancies such as basal cell carcinoma <10 mm are allowed)
* Pregnancy or breast-feeding or, for women of child-bearing potential, unwillingness to use an acceptable form of birth control
* Chronically active hepatitis B or C
* Current history of drug or alcohol abuse or any active liver disease
* Administration of other IMP within 30 days of screening
* Systemic therapy including anti-HER2 therapy within 2 weeks before enrollment
* Ongoing toxicity > grade 2 from previous standard or investigational therapies, according to National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
* History of cardiac disease (myocardial infarction, arrhythmias requiring therapy, symptomatic valvular disease, cardiomyopathy, or pericarditis)
* Evidence of significant medical condition, ongoing severe disease, or laboratory finding that, in the opinion of the Investigator, makes it undesirable for the patient to participate in the study
* Severe claustrophobia, inability to lie flat or fit into the scanner (e.g., body weight ≥350 lbs [160 kg]), or any other inability to tolerate the PET scan
* Known allergies to any product used in this study or any constituents of GEH121224 (18F) Injection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Specific absorbed dose to the target lesions, specific absorbed dose per organ, and total effective dose of [18F]GEH121224. | 6 months
Change in injection site status following administration of [18F]GEH121224 | Before [18F]GEH121224 administration, immediately after dynamic whole body PET/CT scan and single whole body scans
  The occurrence of post-administration injection site status outside the normal limits will be summarized.
Occurrence of Adverse Events (AEs) following administration of [18F]GEH121224 | 6 months
  An overall summary of AEs, SAEs, and [18F]GEH121224-emergent AEs will be presented, coded using the Medical Dictionary for Regulatory Activities (MedDRA) and summarized by system organ class and preferred term.
Changes in heart rate as beats per minute following administration of [18F]GEH121224 | Baseline, before [18F]GEH121224 administration, immediately after dynamic whole body PET/CT scan and single whole body scans
  The occurrence of post-administration heart rate values outside the normal limits will be summarized.
Changes in blood pressure in mmHg following administration of [18F]GEH121224 | Baseline, before [18F]GEH121224 administration, immediately after dynamic whole body PET/CT scan and single whole body scans
  The occurrence of post-administration blood pressure values outside the normal limits will be summarized.
Changes in temperature as degree C following administration of [18F]GEH121224 | Baseline, before [18F]GEH121224 administration, immediately after dynamic whole body PET/CT scan and single whole body scans
  The occurrence of post-administration body temperature values outside the normal limits will be summarized.
Changes in respiration rate as breaths per minute following administration of [18F]GEH121224 | Baseline, before [18F]GEH121224 administration, immediately after dynamic whole body PET/CT scan and single whole body scans
  The occurrence of post-administration respiration rate values outside the normal limits will be summarized.
Change from baseline in the results of 12-lead electrocardiograms (ECGs) following administration of [18F]GEH121224 | Baseline, before [18F]GEH121224 administration, immediately after single whole body PET/CT scans
  Descriptive statistics will be used to describe the observed values and change from baseline for ECG intervals (PR, QTc, QRS or RR).

SECONDARY OUTCOMES:
Biodistribution | 6 months
  Time-activity curves will be generated and integrated to obtain the cumulated activity in each region, and these values will be used to determine the internal radiation dosimetry using the Medical Internal Radiation Dose (MIRD) schema.
Reproducibility | 6 months
  Variation in the relative standardized uptake values (SUVs) calculated from test and retest [18F]GEH121224 PET images.

CONTACTS AND LOCATIONS:
Overall Officials: Eduard Zhalovaga, MD, PhD, Study Director — GE Healthcare Ltd
Locations (1):
- The University of Texas MD Anderson Cancer Centre, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No